CLINICAL TRIAL: NCT06598241
Title: A Pilot, Post-market, Non-interventional, Prospective, Observational Study of Standard of Care of the Commercially Available Borate-base Bioactive Glass Fiber Matrix (BBGFM) in Treatment of Outpatient Diabetic Foot Ulcer With Chronic Osteomyelitis.
Brief Title: Mirragen Diabetic Foot Ulcer Study
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00000049
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Foot Ulcer; Osteomyelitis Chronic
Keywords: Glass fiber matrix
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic Foot Ulcer Treatment Group: Male or female between ≥ 18 years and ≤ 80 years of age that are scheduled to receive treatment of the commercially available borate-based bioactive glass fiber matrix will be enrolled in the study
  Interventions: Device: Borate-base Bioactive Glass Fiber Matrix (BBGFM)

INTERVENTIONS:
Device: Borate-base Bioactive Glass Fiber Matrix (BBGFM) — Bioactive glass materials are biocompatible water-soluble inorganic ceramic materials that release their constituent ions when immersed in body fluids.

SUMMARY:
This study is being done to collect data from treatment of patients who have diabetes with non-healing foot wounds and are being treated with a resorbable and biocompatible borate-based bioactive glass fiber matrix. A borate-based bioactive glass fiber matrix is used to cover the ulcer for wound management. The primary objective of this study is to evaluate the safety and efficacy of the borate-based bioactive glass fiber matrix in the treatment of diabetic foot ulcers in a real-world setting. The secondary objective is to evaluate the clinical and financial benefits in terms of quality of healing, pain, and treatment cost.

DETAILED DESCRIPTION:
While participants are taking part in this study, they will be asked to attend approximately 12 weekly visits, or until the ulcer has healed. After the ulcer has healed there will be two follow up visits for confirmation, these visits are two weeks apart. Visits with the researchers and/or study staff will last for 16 weeks or less. Participants will continue and complete regular follow-up visit with their treating doctor while participating in this study.

The purpose of this study is to collect information about the product safety and efficacy of real-world scenarios on treating diabetic foot ulcers. The data that will be collected will help understand long-term risk and benefit from a real-world population.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has signed the informed consent form
2. Subject is male or female aged between ≥ 18 or ≤ 80
3. Subject scheduled to receive borate-based bioactive glass fiber matrix in treatment of index diabetic foot ulcer
4. Index ulcer has not received an application of BBFGM previously
5. Subjects with insurance coverage for BBGFM
6. Subject has documented Type 1 or Type 2 diabetes with an HbA1c less than or equal to 12.0% within 90 days of enrollment.
7. The subject is under the care of Physician for the management of Diabetes Mellitus
8. Subject must have a wound present anatomically on the foot as defined by beginning below the malleoli of the ankle, dorsal surface, plantar surface, inter digital, heel, lateral or medial surface of the foot
9. Subject index ulcers must be ≥ 0.5 cm2 and ≤ 8.0 cm2
10. Index ulcer has been present for greater than 4 weeks prior to enrollment and less than 2-years, as of the date the subject receives the BBGFM
11. The BBGFM will be applied in an outpatient setting
12. Subject has an ulcer with a Wagner Grade 2 or 3 classification Wagner Grade 2: Deep ulcer extended to ligament, tendon, joint capsule, bone, or deep fascia without abscess or osteomyelitis Wagner Grade 3: Ulcers extend to the deep tissue and have either associated soft tissue abscess or osteomyelitis If Wagner Grade 3 Ulcer with chronic osteomyelitis, that can be debrided in an outpatient setting, in the opinion of the investigator

    1. Exposed or palpable bone in the reference ulcer, that can be surgically excised in an outpatient clinic setting, using local anesthetic, at the screening or randomization visit
    2. Less than a 1cm margin of peri-ulcer tissue of the reference ulcer, requiring surgical debridement, at the screening and randomization visit

    Wagner Grade 3 subjects must have osteomyelitis diagnosed by:

    X-ray: suggestive or positive for changes consistent with chronic osteomyelitis or Positive probe to bone (PTB) test or Strong clinical suspicion, in the opinion of the Investigator, in the presence of osteomyelitis in the index wound
13. Subject does not require a surgical debridement in the operating room
14. Subjects without active cellulitis at the index ulcer
15. Subject or responsible caregiver is willing to comply with the dressing treatment and study visits
16. Subject is willing to utilize the offloading device to offload wound
17. If female, subjects must have been practicing adequate contraception (abstinence, barrier method, hormonal, or IUD). Must agree to using an accepted and effective form of birth control during the study.
18. Subject has adequate circulation to the affected extremity, as demonstrated by at least ONE of the following tests within 60 days (about 2 months) prior to enrollment:

A.Ankle-Brachial Index (ABI) of study leg(s) of ≥0.7 to ≤1.3 in conjunction with doppler arterial waveforms, which are triphasic or biphasic at the ankle of affected leg Or B.Toe brachial Index (TBI) of ≥ 0.50 OR C.Great Toe Pressure 50mmHg OR D.Dorsum transcutaneous oxygen test (TcPO2) of study leg(s) of ≥40mmHg on the dorsum of the affected foot OR E.Palpable pulses

Exclusion Criteria:

1. Subject is unwilling to sign informed consent
2. Subjects who cannot obtain insurance coverage for BBFGM
3. The BBFGM cannot be applied in an outpatient setting
4. Index ulcer has previously received an application of BBFGM
5. Subject has a major contralateral amputation of lower extremity, specifically transmetatarsal amputation or more proximal amputation
6. Subject index ulcer has a known history of borate-base bioactive glass fiber matrix application
7. Subject is pregnant or breast-feeding.
8. Subject index ulcer associated with carcinoma.
9. Subject has active Charcot Neuroarthropathy
10. Subject requires extensive soft tissue and bone debridement in the operating room
11. Subject has a life expectancy of less than six months as assessed by the investigator.
12. Subject not in reasonable metabolic control in the judgment of the investigator
13. Subject with a known history of poor compliance with medical treatments
14. Subject currently undergoing cancer treatment
15. Subject has been on oral steroid use of <7.5 mg daily for greater than seven consecutive days in 30 days before screening
16. Subject is taking parenteral corticosteroids or any cytotoxic agents for seven consecutive days in the period of 30 days before screening
17. The subject has malignancy or a history of cancer, other than non-melanoma skin cancer, in five years before screening
18. Subject has been diagnosed or had medical history with at least one of the following diseases: cancer, lupus, vasculitis, sickle cell, fibromyalgia, acquired immunodeficiency syndrome (AIDS) or HIV, uncontrolled rheumatoid arthritis, stage renal disease.
19. Subject currently receiving radiation therapy or chemotherapy.
20. Patient currently on dialysis or planning to start dialysis.
21. Presence of any condition that is likely to impair understanding of or compliance with the study protocol in the judgment of the Investigator
22. Subject is unable to sustain off-loading as defined by the protocol
23. Subject index ulcer that cannot be offload by an offloading device
24. Subject index ulcer with acute osteomyelitis, as per no bony changes on x-ray and/or presence of acute cellulitis at the index ulcer
25. Subject is anticipated to use Negative Pressure Wound Therapy (NPWT) on the index ulcer during the study
26. Subjects who are permanently non-ambulatory (i.e. wheelchair bound)
27. The subject is a woman of child-bearing potential who is unwilling to avoid pregnancy or use an appropriate form of birth control (adequate birth control methods are defined as: topical, oral, implantable, or injectable contraceptives; spermicide in conjunction with a barrier such as a condom or diaphragm; IUD; or surgical sterilization of partner)
28. Subject has an allergy to primary or secondary dressing materials used in this trial
29. In the opinion of the Investigator the subject is not appropriate for inclusion in the trial, e.g., undergoing surgical treatments listed in the protocol or subject currently has sepsis, i.e., life threatening organ dysfunction caused by a dysregulated host response to infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled to receive treatment of commercially available borate-based bioactive glass fiber matrix (BBGFM) at the Medical Arts and Research Center (MARC) and Texas Diabetes Institute (TDI) will be considered potential subjects and will be pre-screened.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Complete Wound Closure | Week 12
  Number of patients to achieve complete wound closure. Complete wound closure is defined as skin re-epithelialization without drainage or dressing requirements confirmed at 2 consecutive study visits 2 weeks apart.

SECONDARY OUTCOMES:
60% Reduction in wound size | Baseline to 12 weeks
  Percentage of subjects achieving greater than or equal to 60 % reduction in wound area and depth from enrollment visit to 12 weeks, measured weekly with standard ruler and iPhone "Measure" app
Pain level using Visual Analog Scale | Baseline to 12 weeks
  Change in pain levels during trial, using the Visual Analog Scale which measure pain on range of 0 to 10, zero being no pain and 10 being the most severe pain.
Change in Lower Extremity Function Scale (LEFS ) | Baseline to 12 weeks
  The Lower Extremity Functional Scale (LEFS) is a 20-item questionnaire that measures a person's disability in activities related to their lower extremities. The scale is scored on a scale of 0 to 80, with higher scores indicating less disability.
Number of Adverse Events related to BBGFM | Baseline to 12 weeks
  Mean number of adverse events experienced by participants related to the treatment
Number of subjects with either cellulitis, infection and/or osteomyelitis | Baseline to 12 weeks
  Total number of subjects that experience any of these infections during study enrollment
Timing to achieve 100% granulation coverage of wound surface | Baseline to 12 weeks
  Number of weeks to achieve complete granulation coverage of ulcer
Number of Applications to achieve 100% granulation coverage of wound surface | Baseline to 12 weeks
  Average number of borate-based bioactive glass fiber matrix applications
Hospitalization rate for wound related events | Baseline to 12 weeks
  Number of participants hospitalized for wound related events during study
Number of Amputations | Baseline to 12 weeks
  Number of subjects requiring amputations during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Cyaandi R Dove, DPM, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- UT Health Medical Arts and Research Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will ensure all mechanisms used to share data will include proper plans and safeguards for the protection of privacy, confidentiality, and security for data dissemination and reuse (e.g., all data will be thoroughly de-identified and will not be traceable to a specific study participant). Data will be shared when accepted for publication in a peer-review journal
Supporting Information: Study Protocol, SAP
Time Frame: At the time of publication in a peer-review journal